CLINICAL TRIAL: NCT03002480
Title: Individualizing Bypassing Agent Therapy Utilizing TEG in Hemophilia Patients with Inhibitors
Brief Title: Individualizing Hemophilia Bypassing Agent Therapy Utilizing Thromboelastography
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never opened.
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Guy Young, Director of Thrombosis and Hemostasis, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-16-00501
Record Dates: First submitted 2016-12-19; First posted 2016-12-23 (Estimated); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Hemophilia a with Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Severe Hemophilia A subjects w/ inhibitors (Other): Males age 4-70 years diagnosed with severe hemophilia A with inhibitors who are currently treated with prophylaxis or on-demand treatment will be enrolled.
  Interventions: Other: Thromboelastography-Guided Treatment Regimen

INTERVENTIONS:
Other: Thromboelastography-Guided Treatment Regimen — The thromboelastograph (TEG) will be used to determine the "best" bypassing agent for the management of subjects with severe hemophilia A with inhibitors. Patients will be assigned that bypassing agent and dose for the treatment of their bleeding episodes and subsequently will be followed for a period of 6 months to determine their annual bleeding rate.

SUMMARY:
This pilot study will investigate the use of thromboelastograph (TEG) to determine the primary bypassing agent for the management of bleeding in children and adults severe hemophilia A patients with inhibitors.

The study will evaluate the TEG profile for each of the available bypassing agents (FEIBA and rFVIIa) in each participating patient, which will then determine which agent provides the most robust clot formation as measured by the TEG. This study will consist of screening visit and 2-4 pharmacokinetic studies to determine the "best" bypassing agent based on the TEG results. Patients will then be assigned that bypassing agent and dose for the treatment of their bleeding episodes (Prophylaxis or On-demand). Each patient will be then followed for a period of 6 months to monitor short-term safety of those patients whose bypassing agent was modified.

DETAILED DESCRIPTION:
Currently, there are no laboratory assays that can assess the pharmaceutical activity of the available agents known collectively as bypassing agents, which negatively impacts the treating physician's ability to manage these patients, leaving decisions on the dosing regimen to trial and error. Both agents, FEIBA and recombinant activated factor VII (rFVIIa), are approved for the treatment of bleeding in inhibitor patients with recommended dosing regimens that are based on clinical trials. However, a significant amount of "experimenting" with other dosing regimens is used by physicians and patients.

The goal of this project is to demonstrate that TEG is an excellent biomarker for predicting, managing and individualizing the treatment with FEIBA and rFVIIa of this rare and difficult to treat patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Males, 4-60 years old, inclusive on Prophylaxis or On-Demand treatment
2. Diagnosis of Hemophilia with active titer inhibitors (> 0.6 BU)
3. Willing to alter their treatment regimen per study protocol

Exclusion Criteria:

1. Bleeding disorder(s) other than hemophilia A with inhibitors
2. Thrombocytopenia (platelet count <100,000K/µL)
3. Any concurrent clinically significant major disease that, in the opinion of the investigator, would make the subject unsuitable for enrollment
4. Participation within the past 30 days in a clinical study involving investigational drugs
5. Planned major surgery within 30 days prior to screening or during the study period

Ages: 4 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Elastic properties of a forming clot using thromboelastograph to determine best bypassing agent | 6 months
  This study will assess the feasibility of TEG-guided individualization of bypassing agent treatment of bleeding for severe hemophilia A patients with inhibitors.

SECONDARY OUTCOMES:
Thrombin generation assay measuring the formation of thrombin during clot formation | 6 months
  Thrombin generation assays will be performed to provide additional evidence supporting the TEG-guided individualization of bypassing agent treatment.
Number of participants with treatment-related adverse events | 1 year
  The study will monitor short-term safety of patients whose bypassing agent treatment has been modified.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Young, MD, Principal Investigator — Children's Hospital Los Angeles

IPD SHARING:
Plan to Share IPD: No